CLINICAL TRIAL: NCT00568776
Title: A Randomized, Double-Blind, Placebo-Controlled, Dose-Ranging, Safety and Efficacy Study of Oral ELND005 (AZD-103) in Alzheimer's Disease
Brief Title: ELND005 in Patients With Mild to Moderate Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: OPKO Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ELND005-AD201
Record Dates: First submitted 2007-12-04; First posted 2007-12-06 (Estimated); Results first posted 2012-03-29 (Estimated); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — scyllitol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Placebo Comparator)
  Interventions: Drug: Placebo Control
- 2 (Active Comparator)
  Interventions: Drug: ELND005
- 3 (Active Comparator)
  Interventions: Drug: ELND005
- 4 (Active Comparator)
  Interventions: Drug: ELND005

INTERVENTIONS:
Drug: Placebo Control — ELND005 matched placebo capsules for oral administration, bid for 78 weeks
  Other Names: scyllo-inositol
  Arms: 1
Drug: ELND005 — ELND005 capsules for oral administration at a dose of 2000 mg bid for 78 weeks
  Arms: 4
Drug: ELND005 — ELND005 capsules for oral administration at a dose of 250 mg bid for 78 weeks
  Other Names: scyllo-inositol
  Arms: 2
Drug: ELND005 — ELND005 capsules for oral administration at a dose of 1000 mg bid for 78 weeks
  Other Names: scyllo-inositol
  Arms: 3

SUMMARY:
The purpose of this study is to evaluate the dose-related safety and efficacy of multiple oral dosages of ELND005 as treatment for Alzheimer's disease (AD).

DETAILED DESCRIPTION:
ELND005 (formerly known as AZD-103), scyllo-inositol, is being investigated as an orally administered treatment for AD. ELND005 may prevent or inhibit the build up of amyloid protein in the brains of AD patients.

This is a randomized, double-blind, placebo-controlled, dose-ranging, safety and efficacy study of oral ELND005 in male and female participants aged 50-85 years with mild to moderate AD. Approximately 340 patients will be enrolled into the study at approximately 65 study sites. Patients will be randomized to receive either ELND005 or placebo. Each patient's participation will last approximately 18 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of probable AD
* Age 50 to 85 years, inclusive
* Mini-Mental Status Exam (MMSE) score of 16-26, inclusive
* Brain magnetic resonance imaging (MRI) scan consistent with the diagnosis of AD
* Fluency in English, French, or Spanish
* Stable doses of medications (cholinesterase inhibitors and memantine allowed)
* Caregiver is able to attend all study visits

Exclusion Criteria:

* Significant neurological disease other than AD
* Major psychiatric disorder
* Significant medical illness
* History of stroke or seizure
* History of a heart attack within the last 2 years
* Prior treatment with certain experimental medicines
* Presence of pacemakers or foreign metal objects in the eyes, skin, or body that would prevent patient from having MRI scan

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 353 (Actual)
Dates: Start 2007-12; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (62):
- United States (50):
  - Banner Alzheimer's Institute, Phoenix, Arizona
  - Sun Health Research Institute, Sun City, Arizona
  - University of Arizona, Health Sciences Center, Dept. of Neurology, Tucson, Arizona
  - Margolin Brain Institute, Fresno, California
  - Collaborative NeuroScience Network, Inc., Garden Grove, California
  - UCLA Alzheimer's Disease Center, Dept. of Neurology, Los Angeles, California
  - UC Irvine Medical Center, Orange, California
  - UCSF Medical Center, Dept. of Neurology, San Francisco, California
  - Yale University School of Medicine, Alzheimer's Disease Research Unit, New Haven, Connecticut
  - Georgetown University Medical Center, Dept. of Neurology, Washington D.C., District of Columbia
  - Brain Matters Research, Inc., Delray Beach, Florida
  - Sunrise Clinical Research, Inc, Hollywood, Florida
  - Miami Jewish Home and Hospital For The Aged, Miami, Florida
  - Avision Research Associates, LLC, Miami, Florida
  - Compass Research, LLC, Orlando, Florida
  - Roskamp Institute, Sarasota, Florida
  - Neurology Clinical Research, Inc., Sunrise, Florida
  - University of South Florida Suncoast Alzheimer's and Gerontology Center, Tampa, Florida
  - Premiere Research Institute, West Palm Beach, Florida
  - Emory University, Dept. of Neurology, Atlanta, Georgia
  - Dekalb Neurology Associates, LLC, Decatur, Georgia
  - Department of Neurology - Indiana University Medical Center, Indianapolis, Indiana
  - University of Kansas Medical Center, Department of Neurology, Kansas City, Kansas
  - Innovative Clinical Concepts, Paducah, Kentucky
  - Brigham and Women's Hospital, Dept. of Neurology, Boston, Massachusetts
  - University of Michigan, Taubman Health Care Center, Dept. of Neurology, Ann Arbor, Michigan
  - University of Nevada School of Medicine, Las Vegas, Nevada
  - Comprehensive Clinical Research, Berlin, New Jersey
  - The Memory Enhancement Center of America, Inc., Eatontown, New Jersey
  - Global Medical Institutes, Princeton, New Jersey
  - Albuquerque Neuroscience, Inc., Albuquerque, New Mexico
  - Upstate Clinical Research, LLC, Albany, New York
  - Neurological Associates of Albany, PC, Albany, New York
  - Mount Sinai Medical Center, New York, New York
  - Columbia University Sergievsky Center, New York, New York
  - AD-CARE, Monroe Community Hospital, Rochester, New York
  - Raleigh Neurology Associates, Raleigh, North Carolina
  - Neurology & Neuroscience Center of Ohio, Toledo, Ohio
  - Medford Neurological and Spine Clinic, Medford, Oregon
  - Summit Research Newtwork, Inc., Portland, Oregon
  - Abington Neurological Associates, Inc., Abington, Pennsylvania
  - The Clinical Trial Center, LLC, Jenkintown, Pennsylvania
  - University of Pittsburgh Alzheimer Disease Research Clinic, Pittsburgh, Pennsylvania
  - Butler Hospital, Memory and Aging Center, Providence, Rhode Island
  - Alliance for Neuro Research, LLC dba Absher Neurology, PA, Greenville, South Carolina
  - Radiant Research San Antonio, San Antonio, Texas
  - University of Utah, Dept. of Neurology, Salt Lake City, Utah
  - Clinical Neuroscience Research Associates, Inc-The Memory Clinic, Bennington, Vermont
  - University of Vermont Medical Center, Fletcher Allen Health Care, Dept. of Neurology, Burlington, Vermont
  - University of Virginia Health System, Charlottesville, Virginia
- Canada (12):
  - Glenrose Rehabilitation Hospital, Edmonton, Alberta
  - University of British Columbia Hospital, Division of Neurology, Vancouver, British Columbia
  - Hotel Dieu Hospital, Kingston, Ontario
  - Saint Joseph's Health Care London, Saint Joseph's Hospital, Dept. of Cognitive Neurology, London, Ontario
  - Parkwood Hospital, London, Ontario
  - Sisters of Charity of Ottawa Health Service, Ottawa, Ontario
  - Kawartha Regional Memory Clinic, Peterborough, Ontario
  - Toronto Memory Program, Toronto, Ontario
  - Whitby Mental Health Memory Clinic, Toronto, Ontario
  - Gerontion Research, Inc., Toronto, Ontario
  - Neuro-Rive-Sud Memory Clinic, Greenfield Park, Quebec
  - Recherche Clinique de Neurologie (Hospital Maisonneuve Rosemont), Montreal, Quebec

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo BID; ELND005 250 mg BID; ELND005 1000 mg BID; ELND005 2000 mg BID: oral administration for 78 weeks
Period: Overall Study
Arm/Group | Placebo BID | ELND005 250 mg BID | ELND005 1000 mg BID | ELND005 2000 mg BID
Started | 83 (One randomized patient withdrew consent and did not receive placebo) | 88 (One randomized patient withdrew consent and did not receive ELND005 250 mg BID) | 89 (41 patients withdrawn per interim safety review (sponsors decision); excluded in efficacy analysis.) | 91 (42 patients withdrawn per interim safety review (sponsors decision); excluded in efficacy analysis.)
Completed | 53 | 52 | 15 | 19
Not Completed | 30 | 36 | 74 | 72
Not completed — Adverse Event | 8 | 8 | 10 | 8
Not completed — Death | 0 | 1 | 4 | 3
Not completed — Physician Decision | 0 | 2 | 0 | 0
Not completed — Lack of Efficacy | 2 | 2 | 2 | 4
Not completed — Lost to Follow-up | 1 | 1 | 1 | 1
Not completed — Protocol Violation | 1 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 13 | 15 | 13 | 7
Not completed — Loss of Caregiver | 0 | 2 | 1 | 2
Not completed — Sponsor Decision | 2 | 2 | 41 | 42
Not completed — Miscellaeneous | 3 | 3 | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo BID | ELND005 250 mg BID | ELND005 1000 mg BID | ELND005 2000 mg BID | Total
Number analyzed (Participants) | 83 | 88 | 89 | 91 | 351
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.4 (7.83) | 73.4 (7.26) | 73.4 (7.56) | 72.2 (8.20) | 73.1 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 51 | 48 | 51 | 197
  Male | 36 | 37 | 41 | 40 | 154
Region of Enrollment [Number; unit: patients]
  United States | 68 | 75 | 71 | 75 | 289
  Canada | 15 | 13 | 18 | 16 | 62

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 78 in Neuropsychological Test Battery (NTB) Z-score (Full Analysis Set; FAS)
Description: The NTB assessment is comprised of 9 instruments that measure cognition and executive function. Three of these tests measure immediate memory, next three measure delayed memory, and remaining three assess executive function. The total score is a weighted mean of the nine tests, referred to as the Z-score. Typically, scores range from -3 and 3, with lower scores suggesting greater cognitive impairment.
Time Frame: Baseline and 78 weeks
Population: Full Analysis Set (FAS): all randomized patients who received at least one dose of study drug and completed the baseline visit and at least one post-baseline visit.
Measure: Mean (Standard Error); unit: Scores on a Scale
Arm/Group | Placebo BID | ELND005 250 mg BID | ELND005 1000 mg BID | ELND005 2000 mg BID
Number analyzed (Participants) | 82 | 84 | 0 | 0
Scores on a Scale | -0.383 (0.075) | -0.350 (0.074) |  |
Statistical Analysis 1: Comparison: Placebo BID vs ELND005 250 mg BID; Test type: Superiority or Other; p = 0.71, Mixed Models Analysis; Mean Difference (Final Values) = 0.03, 95% CI 2-sided [-0.14 to 0.21], Standard Error of Mean 0.09

2. Secondary Outcome: Change in Alzheimer's Disease Assessment Scale - Cognitive Subscale (ADAS-Cog) Score From Baseline to Week 78 (Full Analysis Set; FAS)
Description: The ADAS-Cog primarily measures cognitive ability. The version used in this study was comprised of 12 items with scores ranging from 0 to 75. Higher scores suggest greater cognitive impairment.
Time Frame: Baseline and 78 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Scores on a Scale
Arm/Group | Placebo BID | ELND005 250 mg BID | ELND005 1000 mg BID | ELND005 2000 mg BID
Number analyzed (Participants) | 82 | 84 | 0 | 0
Scores on a Scale | -8.239 (1.531) | -10.796 (1.540) |  |
Statistical Analysis 1: Comparison: Placebo BID vs ELND005 250 mg BID; Test type: Superiority or Other; p = 0.18, Mixed Models Analysis; Mean Difference (Final Values) = -2.56, 95% CI 2-sided [-6.33 to 1.22], Standard Error of Mean 1.90

3. Primary Outcome: Additional Analysis of Primary Outcome Measure: Change From Baseline to Week 78 in Neuropsychological Test Battery (NTB) Z-score (Per Protocol Set; PPS)
Description: as for outcome 1
Time Frame: Baseline and 78 weeks
Population: Per Protocol Set (PPS): all randomized patients who received at least one dose of ELND005 250 mg or placebo, completed all scheduled visits up to Week 78, were at least 80% compliant with study drug, and met all inclusion/exclusion criteria.
Measure: Mean (Standard Error); unit: Scores on a Scale
Arm/Group | Placebo BID | ELND005 250 mg BID | ELND005 1000 mg BID | ELND005 2000 mg BID
Number analyzed (Participants) | 47 | 49 | 0 | 0
Scores on a Scale | -0.369 (0.093) | -0.222 (0.095) |  |
Statistical Analysis 1: Comparison: Placebo BID vs ELND005 250 mg BID; Test type: Superiority or Other; p = 0.17, Mixed Models Analysis; Mean Difference (Final Values) = 0.15, 95% CI 2-sided [-0.06 to 0.36], Standard Error of Mean 0.11

4. Primary Outcome: Change From Baseline to Week 78 in Alzheimer's Disease Cooperative Study - Activities of Daily Living (ADCS-ADL) Score (Full Analysis Set; FAS)
Description: The ADCS-ADL is a 23-item scale that measures a subject's functional abilities as assessed by the subject's caregiver. This scale ranges from 0 to 78, with lower scores suggesting greater functional impairment.
Time Frame: Baseline and 78 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Scores on a Scale
Arm/Group | Placebo BID | ELND005 250 mg BID | ELND005 1000 mg BID | ELND005 2000 mg BID
Number analyzed (Participants) | 82 | 84 | 0 | 0
Scores on a Scale | -9.467 (1.641) | -10.861 (1.604) |  |
Statistical Analysis 1: Comparison: Placebo BID vs ELND005 250 mg BID; Test type: Superiority or Other; p = 0.49, Mixed Models Analysis; Mean Difference (Final Values) = -1.39, 95% CI 2-sided [-5.41 to 2.62], Standard Error of Mean 2.03

5. Primary Outcome: Additional Analysis of Primary Outcome Measure: Change From Baseline to Week 78 in Alzheimer's Disease Cooperative Study - Activities of Daily Living (ADCS-ADL) Score (Per Protocol Set; PPS)
Description: as for outcome 4
Time Frame: Baseline and 78 weeks
Population: as for outcome 3
Measure: Mean (Standard Error); unit: Scores on a Scale
Arm/Group | Placebo BID | ELND005 250 mg BID | ELND005 1000 mg BID | ELND005 2000 mg BID
Number analyzed (Participants) | 47 | 49 | 0 | 0
Scores on a Scale | -9.635 (1.779) | -8.987 (1.760) |  |
Statistical Analysis 1: Comparison: Placebo BID vs ELND005 250 mg BID; Test type: Superiority or Other; p = 0.77, Mixed Models Analysis; Mean Difference (Final Values) = 0.65, 95% CI 2-sided [-3.73 to 5.03], Standard Error of Mean 2.20

6. Secondary Outcome: Change in Clinical Dementia Rating - Sum of Boxes (CDR-SB) Score From Baseline to Week 78 (Full Analysis Set; FAS)
Description: The CDR-SB consists of 6 items; 3 measuring cognitive ability and 3 measuring functional ability. The score for each of the six items range from 0 to 3; hence the total score is between 0 and 18. Higher scores suggest greater cognitive impairment.
Time Frame: Baseline and 78 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Scores on a Scale
Arm/Group | Placebo BID | ELND005 250 mg BID | ELND005 1000 mg BID | ELND005 2000 mg BID
Number analyzed (Participants) | 82 | 84 | 0 | 0
Scores on a Scale | -2.742 (0.363) | -2.452 (0.357) |  |
Statistical Analysis 1: Comparison: Placebo BID vs ELND005 250 mg BID; Test type: Superiority or Other; p = 0.54, Mixed Models Analysis; Mean Difference (Final Values) = 0.29, 95% CI 2-sided [-0.63 to 1.21], Standard Error of Mean 0.47

7. Secondary Outcome: Change in Neuropsychiatric Inventory (NPI) Score From Baseline to Week 78 (Full Analysis Set; FAS)
Description: The NPI is used to obtain information on the presence of severity of neuropsychological symptoms, and was specifically designed for use in Alzheimer's disease subjects. The scale consists of 12 items with each item having outcomes from 0 to 12; hence the total score ranges from 0 to 144. Higher scores suggest greater psychiatric impairment.
Time Frame: Baseline and 78 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Scores on a Scale
Arm/Group | Placebo BID | ELND005 250 mg BID | ELND005 1000 mg BID | ELND005 2000 mg BID
Number analyzed (Participants) | 82 | 84 | 0 | 0
Scores on a Scale | -6.132 (1.851) | -5.116 (1.814) |  |
Statistical Analysis 1: Comparison: Placebo BID vs ELND005 250 mg BID; Test type: Superiority or Other; p = 0.65, Mixed Models Analysis; Mean Difference (Final Values) = 1.02, 95% CI 2-sided [-3.43 to 5.46], Standard Error of Mean 2.24

ADVERSE EVENTS:
Time Frame: Reported adverse events include events starting at or after Screening to Week 84
Description: For all adverse event (AE) summaries, if a patient had more than one AE within a preferred term the patient was counted only once, at the maximum severity and with the closest relationship to study drug. If a patient had more than one AE within a system organ class (SOC), the patient was similarly counted once when reporting results for that SOC.
Arm/Group | Placebo BID | ELND005 250 mg BID | ELND005 1000 mg BID | ELND005 2000 mg BID
Serious Adverse Events (participants affected / at risk) | 11/83 | 19/88 | 20/89 | 21/91
Other Adverse Events (participants affected / at risk) | 48/83 | 46/88 | 45/89 | 57/91
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo BID (N=83) | ELND005 250 mg BID (N=88) | ELND005 1000 mg BID (N=89) | ELND005 2000 mg BID (N=91)
Angina Unstable (Cardiac disorders) | 1 | 0 | 0 | 0
Atrial Fribrillation (Cardiac disorders) | 1 | 1 | 1 | 1
Atrial Futter (Cardiac disorders) | 1 | 1 | 0 | 0
Cardiac Arrest (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiac Failure Congestive (Cardiac disorders) | 0 | 0 | 0 | 2
Coronary Artery Occlusion (Cardiac disorders) | 0 | 1 | 0 | 0
Myocardial Infarction (Cardiac disorders) | 1 | 1 | 0 | 0
Supraventricular Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Glaucoma (Eye disorders) | 1 | 0 | 0 | 0
Retinal Vein Occlusion (Eye disorders) | 1 | 0 | 0 | 0
Vitreous Haemorrhage (Eye disorders) | 1 | 0 | 0 | 0
Gastric Ulcer Haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastritis Hemorrhagic (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Hypothermia (General disorders) | 1 | 0 | 0 | 0
Sudden Death (General disorders) | 0 | 0 | 1 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Arthritis Bacterial (Infections and infestations) | 0 | 0 | 0 | 1
Bacterial Sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Kidney Infection (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 2 | 3
Pneumonia Bacterial (Infections and infestations) | 0 | 0 | 1 | 0
Staphylococcal Infection (Infections and infestations) | 0 | 0 | 0 | 1
Urinary Tract Infection (Infections and infestations) | 1 | 0 | 0 | 3
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 1
Viral Infection (Infections and infestations) | 0 | 1 | 0 | 0
Accidental Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Compression Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Hip Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Jaw Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Multiple Fractures (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Post Procedural Haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Postoperative Ileus (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Subdural Hematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Electrocardiogram Change (Investigations) | 0 | 0 | 1 | 0
Hepatic Enzyme Increased (Investigations) | 0 | 0 | 1 | 0
Lipase Increased (Investigations) | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 1 | 2 | 2
Failure to Thrive (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Mobility Decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3 | 0 | 0
Breast Cancer In Situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Colorectal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 2
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Squamous Cell Carcinoma of Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Carotid Artery Occlusion (Nervous system disorders) | 1 | 0 | 0 | 0
Cerebral Hemorrhage (Nervous system disorders) | 0 | 1 | 0 | 0
Cerebrovascular Accident (Nervous system disorders) | 0 | 0 | 1 | 1
Dementia Alzheimer's Type (Nervous system disorders) | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 1
Haemorrhagic Stroke (Nervous system disorders) | 1 | 0 | 0 | 0
Ischaemic Cerebral Infarction (Nervous system disorders) | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 1
Transient Ischaemic Attack (Nervous system disorders) | 0 | 0 | 1 | 0
Acute Psychosis (Psychiatric disorders) | 0 | 0 | 0 | 1
Agitation (Psychiatric disorders) | 0 | 1 | 1 | 0
Confusional State (Psychiatric disorders) | 0 | 0 | 1 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 1 | 0
Mental Status Changes (Psychiatric disorders) | 1 | 0 | 0 | 0
Psychotic Disorder (Psychiatric disorders) | 0 | 0 | 1 | 1
Renal Failure Acute (Renal and urinary disorders) | 0 | 0 | 2 | 0
Urinary Retention (Renal and urinary disorders) | 0 | 0 | 1 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Aortic Thrombosis (Vascular disorders) | 0 | 1 | 0 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 1 | 0 | 0
Haemorrhagic Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo BID (N=83) | ELND005 250 mg BID (N=88) | ELND005 1000 mg BID (N=89) | ELND005 2000 mg BID (N=91)
Diarrhoea (Gastrointestinal disorders) | 6 | 9 | 8 | 12
Nausea (Gastrointestinal disorders) | 4 | 8 | 3 | 14
Vomiting (Gastrointestinal disorders) | 3 | 5 | 3 | 8
Fatigue (General disorders) | 4 | 6 | 6 | 7
Urinary Tract Infection (Infections and infestations) | 7 | 12 | 4 | 11
Fall (Injury, poisoning and procedural complications) | 5 | 11 | 10 | 14
Dizziness (Nervous system disorders) | 7 | 4 | 6 | 11
Headache (Nervous system disorders) | 12 | 4 | 11 | 8
Agitation (Psychiatric disorders) | 5 | 4 | 9 | 6
Confusional State (Psychiatric disorders) | 3 | 7 | 4 | 4
Depression (Psychiatric disorders) | 4 | 10 | 4 | 12
Insomnia (Psychiatric disorders) | 5 | 3 | 2 | 8
Upper Respiratory Tract Infection (Infections and infestations) | 5 | 9 | 3 | 3

LIMITATIONS AND CAVEATS:
The two high dose groups of ELND005 were discontinued before study end, so the efficacy analysis was based only on placebo and ELND005 250 mg bid groups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator may publish after release of multi-center study publication, or 18 months after database lock of overall study. Sponsor has 60 days to review any proposed publication and request removal of Sponsor's confidential information. Sponsor may request an additional 90 days if filing a patent.